CLINICAL TRIAL: NCT00338260
Title: A Triple-Blind, Parallel Study to Investigate the Effect of Losartan Versus Atenolol on the Reduction of Morbidity and Mortality in Hypertensive Patients With Left Ventricular Hypertrophy
Brief Title: Losartan Intervention For Endpoint Reduction in Hypertension (LIFE) Study (0954-133)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0954-133; 2006_502
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension and Left Ventricular Hypertrophy (Thickening of the Main Pumping Chamber of the Heart)
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0954, /Duration of Treatment : 5 Years
Drug: Comparator : atenolol /Duration of Treatment : 5 Years

SUMMARY:
The LIFE study was conducted from 1995-2001. This study was conducted in 9193 patients with high blood pressure and thickening of the main pumping chamber of the heart. The results showed that after an average treatment time of 4.8 years, treatment that was based on losartan was better than treatment based on atenolol for reducing the risk of having a stroke. The main study results were published in Dahlof et al. Lancet 2002;359:995-1003.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 to 80 years
* Males and females
* Hypertension (160-200/95-115 mm Hg
* ECG evidence of left ventricular hypertrophy

Exclusion Criteria:

* Need for treatment with angiotensin converting enzyme inhibitors, or open- label angiotensin receptor blockers or beta-blockers
* Myocardial infarction or stroke within 6 months

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 1995-06; Primary Completion 2001-09 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Composite of cardiovascular death, fatal and nonfatal stroke, fatal and nonfatal myocardial infarction (heart attack)

SECONDARY OUTCOMES:
cardiovascular death, stroke, myocardial infarction, all-cause mortality, hospitalization for heart failure, new-onset diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Dahlof B, Devereux RB, Kjeldsen SE, Julius S, Beevers G, de Faire U, Fyhrquist F, Ibsen H, Kristiansson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H; LIFE Study Group. Cardiovascular morbidity and mortality in the Losartan Intervention For Endpoint reduction in hypertension study (LIFE): a randomised trial against atenolol. Lancet. 2002 Mar 23;359(9311):995-1003. doi: 10.1016/S0140-6736(02)08089-3. PMID 11937178
- [Background] Lindholm LH, Ibsen H, Dahlof B, Devereux RB, Beevers G, de Faire U, Fyhrquist F, Julius S, Kjeldsen SE, Kristiansson K, Lederballe-Pedersen O, Nieminen MS, Omvik P, Oparil S, Wedel H, Aurup P, Edelman J, Snapinn S; LIFE Study Group. Cardiovascular morbidity and mortality in patients with diabetes in the Losartan Intervention For Endpoint reduction in hypertension study (LIFE): a randomised trial against atenolol. Lancet. 2002 Mar 23;359(9311):1004-10. doi: 10.1016/S0140-6736(02)08090-X. PMID 11937179
- [Background] Devereux RB, Dahlof B, Gerdts E, Boman K, Nieminen MS, Papademetriou V, Rokkedal J, Harris KE, Edelman JM, Wachtell K. Regression of hypertensive left ventricular hypertrophy by losartan compared with atenolol: the Losartan Intervention for Endpoint Reduction in Hypertension (LIFE) trial. Circulation. 2004 Sep 14;110(11):1456-62. doi: 10.1161/01.CIR.0000141573.44737.5A. Epub 2004 Aug 23. PMID 15326072
- [Background] Okin PM, Devereux RB, Jern S, Kjeldsen SE, Julius S, Nieminen MS, Snapinn S, Harris KE, Aurup P, Edelman JM, Dahlof B; Losartan Intervention for Endpoint reduction in hypertension Study Investigations. Regression of electrocardiographic left ventricular hypertrophy by losartan versus atenolol: The Losartan Intervention for Endpoint reduction in Hypertension (LIFE) Study. Circulation. 2003 Aug 12;108(6):684-90. doi: 10.1161/01.CIR.0000083724.28630.C3. Epub 2003 Jul 28. PMID 12885747
- [Background] Wachtell K, Hornestam B, Lehto M, Slotwiner DJ, Gerdts E, Olsen MH, Aurup P, Dahlof B, Ibsen H, Julius S, Kjeldsen SE, Lindholm LH, Nieminen MS, Rokkedal J, Devereux RB. Cardiovascular morbidity and mortality in hypertensive patients with a history of atrial fibrillation: The Losartan Intervention For End Point Reduction in Hypertension (LIFE) study. J Am Coll Cardiol. 2005 Mar 1;45(5):705-11. doi: 10.1016/j.jacc.2004.06.080. PMID 15734614
- [Background] Ibsen H, Wachtell K, Olsen MH, Borch-Johnsen K, Lindholm LH, Mogensen CE, Dahlof B, Devereux RB, de Faire U, Fyhrquist F, Julius S, Kjeldsen SE, Lederballe-Pedersen O, Nieminen MS, Omvik P, Oparil S, Wan Y; LIFE substudy. Does albuminuria predict cardiovascular outcome on treatment with losartan versus atenolol in hypertension with left ventricular hypertrophy? A LIFE substudy. J Hypertens. 2004 Sep;22(9):1805-11. doi: 10.1097/00004872-200409000-00026. PMID 15311110
- [Background] Kjeldsen SE, Dahlof B, Devereux RB, Julius S, Aurup P, Edelman J, Beevers G, de Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Snapinn S, Wedel H; LIFE (Losartan Intervention for Endpoint Reduction) Study Group. Effects of losartan on cardiovascular morbidity and mortality in patients with isolated systolic hypertension and left ventricular hypertrophy: a Losartan Intervention for Endpoint Reduction (LIFE) substudy. JAMA. 2002 Sep 25;288(12):1491-8. doi: 10.1001/jama.288.12.1491. PMID 12243636
- [Background] Lindholm LH, Ibsen H, Borch-Johnsen K, Olsen MH, Wachtell K, Dahlof B, Devereux RB, Beevers G, de Faire U, Fyhrquist F, Julius S, Kjeldsen SE, Kristianson K, Lederballe-Pedersen O, Nieminen MS, Omvik P, Oparil S, Wedel H, Aurup P, Edelman JM, Snapinn S; LIFE study group. Risk of new-onset diabetes in the Losartan Intervention For Endpoint reduction in hypertension study. J Hypertens. 2002 Sep;20(9):1879-86. doi: 10.1097/00004872-200209000-00035. PMID 12195132
- [Background] Devereux RB, Dahlof B, Kjeldsen SE, Julius S, Aurup P, Beevers G, Edelman JM, de Faire U, Fyhrquist F, Helle Berg S, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Snapinn S, Wedel H; LIFE Study Group. Effects of losartan or atenolol in hypertensive patients without clinically evident vascular disease: a substudy of the LIFE randomized trial. Ann Intern Med. 2003 Aug 5;139(3):169-77. doi: 10.7326/0003-4819-139-3-200308050-00006. PMID 12899584
- [Background] Wachtell K, Lehto M, Gerdts E, Olsen MH, Hornestam B, Dahlof B, Ibsen H, Julius S, Kjeldsen SE, Lindholm LH, Nieminen MS, Devereux RB. Angiotensin II receptor blockade reduces new-onset atrial fibrillation and subsequent stroke compared to atenolol: the Losartan Intervention For End Point Reduction in Hypertension (LIFE) study. J Am Coll Cardiol. 2005 Mar 1;45(5):712-9. doi: 10.1016/j.jacc.2004.10.068. PMID 15734615
- [Background] Okin PM, Gerdts E, Kjeldsen SE, Julius S, Edelman JM, Dahlof B, Devereux RB; Losartan Intervention for Endpoint Reduction in Hypertension Study Investigators. Gender differences in regression of electrocardiographic left ventricular hypertrophy during antihypertensive therapy. Hypertension. 2008 Jul;52(1):100-6. doi: 10.1161/HYPERTENSIONAHA.108.110064. Epub 2008 May 26. PMID 18504323
- [Background] Li Z, Dahlof B, Okin PM, Kjeldsen SE, Wachtell K, Ibsen H, Nieminen MS, Jern S, Devereux RB. Left bundle branch block and cardiovascular morbidity and mortality in hypertensive patients with left ventricular hypertrophy: the Losartan Intervention For Endpoint Reduction in Hypertension study. J Hypertens. 2008 Jun;26(6):1244-9. doi: 10.1097/HJH.0b013e3282fcc23c. PMID 18475164
- [Background] Boersma C, Carides GW, Atthobari J, Voors AA, Postma MJ. An economic assessment of losartan-based versus atenolol-based therapy in patients with hypertension and left-ventricular hypertrophy: results from the Losartan Intervention For Endpoint reduction (LIFE) study adapted to The Netherlands. Clin Ther. 2007 May;29(5):963-971. doi: 10.1016/j.clinthera.2007.05.014. PMID 17697915
- [Background] Aurigemma GP, Devereux RB, Wachtell K, Palmieri V, Boman K, Gerdts E, Nieminen MS, Papademetriou V, Dahlof B. Left ventricular mass regression in the LIFE study: effect of previous antihypertensive treatment. Am J Hypertens. 2003 Mar;16(3):180-6. doi: 10.1016/s0895-7061(02)03258-2. PMID 12620695
- [Background] Boman K, Olofsson M, Dahlof B, Gerdts E, Nieminen MS, Papademetriou V, Wachtell K, Devereux RB. Left ventricular structure and function in sedentary and physically active subjects with left ventricular hypertrophy (the LIFE Study). Am J Cardiol. 2005 Jan 15;95(2):280-3. doi: 10.1016/j.amjcard.2004.09.019. PMID 15642571
- [Background] Biederman RW, Doyle M, Young AA, Devereux RB, Kortright E, Perry G, Bella JN, Oparil S, Calhoun D, Pohost GM, Dell'Italia LJ. Marked regional left ventricular heterogeneity in hypertensive left ventricular hypertrophy patients: a losartan intervention for endpoint reduction in hypertension (LIFE) cardiovascular magnetic resonance and echocardiographic substudy. Hypertension. 2008 Aug;52(2):279-86. doi: 10.1161/HYPERTENSIONAHA.108.109819. Epub 2008 Jul 7. PMID 18606908
- [Background] Bella JN, Wachtell K, Palmieri V, Liebson PR, Gerdts E, Ylitalo A, Koren MJ, Pedersen OL, Rokkedal J, Dahlof B, Roman MJ, Devereux RB. Relation of left ventricular geometry and function to systemic hemodynamics in hypertension: the LIFE Study. Losartan Intervention For Endpoint Reduction in Hypertension Study. J Hypertens. 2001 Jan;19(1):127-34. doi: 10.1097/00004872-200101000-00017. PMID 11204292
- [Background] Bella JN, Palmieri V, Wachtell K, Liu JE, Gerdts E, Nieminen MS, Koren MJ, Zabalgoitia M, Wright JT, Dahlof B, Devereux RB. Sex-related difference in regression of left ventricular hypertrophy with antihypertensive treatment: the LIFE study. J Hum Hypertens. 2004 Jun;18(6):411-6. doi: 10.1038/sj.jhh.1001708. PMID 15042116
- [Background] Bang LE, Wiinberg N, Wachtell K, Larsen J, Olsen MH, Tuxen C, Hildebrandt PR, Ibsen H. Losartan versus atenolol on 24-hour ambulatory blood pressure. A LIFE substudy. Blood Press. 2007;16(6):392-7. doi: 10.1080/08037050701642808. PMID 18058457
- [Background] Chinali M, de Simone G, Wachtell K, Gerdts E, Gardin JM, Boman K, Nieminen MS, Papademetriou V, Dahlof B, Devereux RB. Left atrial systolic force in hypertensive patients with left ventricular hypertrophy: the LIFE study. J Hypertens. 2008 Jul;26(7):1472-6. doi: 10.1097/HJH.0b013e3282ff84d7. PMID 18551025
- [Background] Christensen MK, Olsen MH, Wachtell K, Tuxen C, Fossum E, Bang LE, Wiinberg N, Devereux RB, Kjeldsen SE, Hildebrandt P, Rokkedal J, Ibsen H. Does long-term losartan- vs atenolol-based antihypertensive treatment influence collagen markers differently in hypertensive patients? A LIFE substudy. Blood Press. 2006;15(4):198-206. doi: 10.1080/08037050600962968. PMID 17078155
- [Background] Devereux RB, Bella J, Boman K, Gerdts E, Nieminen MS, Rokkedal J, Papademetriou V, Wachtell K, Wright J, Paranicas M, Okin PM, Roman MJ, Smith G, Dahlof B. Echocardiographic left ventricular geometry in hypertensive patients with electrocardiographic left ventricular hypertrophy: The LIFE Study. Blood Press. 2001;10(2):74-82. doi: 10.1080/08037050152112050. PMID 11467763
- [Background] Cicala S, Devereux RB, de Simone G, Wachtell K, Gerdts E, Boman K, Nieminen MS, Papademetriou V, Dahlof B, Okin PM. Electrocardiographic and echocardiographic detection of myocardial infarction in patients with left-ventricular hypertrophy. The LIFE Study. Am J Hypertens. 2007 Jul;20(7):771-6. doi: 10.1016/j.amjhyper.2007.01.021. PMID 17586412
- [Background] de Simone G, Wachtell K, Palmieri V, Hille DA, Beevers G, Dahlof B, de Faire U, Fyhrquist F, Ibsen H, Julius S, Kjeldsen SE, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Devereux RB. Body build and risk of cardiovascular events in hypertension and left ventricular hypertrophy: the LIFE (Losartan Intervention For Endpoint reduction in hypertension) study. Circulation. 2005 Apr 19;111(15):1924-31. doi: 10.1161/01.CIR.0000161799.91577.0A. PMID 15837945
- [Background] Gerdts E, Cramariuc D, de Simone G, Wachtell K, Dahlof B, Devereux RB. Impact of left ventricular geometry on prognosis in hypertensive patients with left ventricular hypertrophy (the LIFE study). Eur J Echocardiogr. 2008 Nov;9(6):809-15. doi: 10.1093/ejechocard/jen155. Epub 2008 May 13. PMID 18490279
- [Background] Franklin SS, Wachtell K, Papademetriou V, Olsen MH, Devereux RB, Fyhrquist F, Ibsen H, Kjeldsen SE, Dahlof B. Cardiovascular morbidity and mortality in hypertensive patients with lower versus higher risk: a LIFE substudy. Hypertension. 2005 Sep;46(3):492-9. doi: 10.1161/01.HYP.0000179604.42845.8d. Epub 2005 Aug 22. PMID 16116047
- [Background] Fossum E, Moan A, Kjeldsen SE, Devereux RB, Julius S, Snapinn SM, Edelman JM, de Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H, Dahlof B; LIFE Study Group. The effect of losartan versus atenolol on cardiovascular morbidity and mortality in patients with hypertension taking aspirin: the Losartan Intervention for Endpoint Reduction in hypertension (LIFE) study. J Am Coll Cardiol. 2005 Sep 6;46(5):770-5. doi: 10.1016/j.jacc.2005.05.060. PMID 16139123
- [Background] Devereux RB, Wachtell K, Gerdts E, Boman K, Nieminen MS, Papademetriou V, Rokkedal J, Harris K, Aurup P, Dahlof B. Prognostic significance of left ventricular mass change during treatment of hypertension. JAMA. 2004 Nov 17;292(19):2350-6. doi: 10.1001/jama.292.19.2350. PMID 15547162
- [Background] Gerdts E, Bjornstad H, Toft S, Devereux RB, Omvik P. Impact of diastolic Doppler indices on exercise capacity in hypertensive patients with electrocardiographic left ventricular hypertrophy (a LIFE substudy). J Hypertens. 2002 Jun;20(6):1223-9. doi: 10.1097/00004872-200206000-00037. PMID 12023695
- [Background] Fossum E, Gleim GW, Kjeldsen SE, Kizer JR, Julius S, Devereux RB, Brady WE, Hille DA, Lyle PA, Dahlof B. The effect of baseline physical activity on cardiovascular outcomes and new-onset diabetes in patients treated for hypertension and left ventricular hypertrophy: the LIFE study. J Intern Med. 2007 Oct;262(4):439-48. doi: 10.1111/j.1365-2796.2007.01808.x. PMID 17875180
- [Background] Fyhrquist F, Dahlof B, Devereux RB, Kjeldsen SE, Julius S, Beevers G, de Faire U, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Hille DA, Lyle PA, Edelman JM, Snapinn SM, Wedel H; LIFE Study Group. Pulse pressure and effects of losartan or atenolol in patients with hypertension and left ventricular hypertrophy. Hypertension. 2005 Apr;45(4):580-5. doi: 10.1161/01.HYP.0000161186.55933.6b. PMID 15790960
- [Background] Devereux RB, Roman MJ, Palmieri V, Okin PM, Boman K, Gerdts E, Nieminen MS, Papademetriou V, Wachtell K, Dahlof B. Left ventricular wall stresses and wall stress-mass-heart rate products in hypertensive patients with electrocardiographic left ventricular hypertrophy: the LIFE study. Losartan Intervention For Endpoint reduction in hypertension. J Hypertens. 2000 Aug;18(8):1129-38. doi: 10.1097/00004872-200018080-00019. PMID 10954006
- [Background] Devereux RB, Lyle PA. Losartan for the treatment of hypertension and left ventricular hypertrophy: the Losartan Intervention For Endpoint reduction in hypertension (LIFE) study. Expert Opin Pharmacother. 2004 Nov;5(11):2311-20. doi: 10.1517/14656566.5.11.2311. PMID 15500378
- [Background] Devereux RB, Palmieri V, Liu JE, Wachtell K, Bella JN, Boman K, Gerdts E, Nieminen MS, Papademetriou V, Dahlof B. Progressive hypertrophy regression with sustained pressure reduction in hypertension: the Losartan Intervention For Endpoint Reduction study. J Hypertens. 2002 Jul;20(7):1445-50. doi: 10.1097/00004872-200207000-00033. PMID 12131543
- [Background] Gerdts E, Oikarinen L, Palmieri V, Otterstad JE, Wachtell K, Boman K, Dahlof B, Devereux RB; Losartan Intervention For Endpoint Reduction in Hypertension (LIFE) Study. Correlates of left atrial size in hypertensive patients with left ventricular hypertrophy: the Losartan Intervention For Endpoint Reduction in Hypertension (LIFE) Study. Hypertension. 2002 Mar 1;39(3):739-43. doi: 10.1161/hy0302.105683. PMID 11897755
- [Background] Devereux RB, de Faire U, Fyhrquist F, Harris KE, Ibsen H, Kjeldsen SE, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H, Hille DA, Dahlof B. Blood pressure reduction and antihypertensive medication use in the losartan intervention for endpoint reduction in hypertension (LIFE) study in patients with hypertension and left ventricular hypertrophy. Curr Med Res Opin. 2007 Feb;23(2):259-70. doi: 10.1185/030079906X162854. PMID 17288679
- [Background] Eijkelkamp WB, Zhang Z, Brenner BM, Cooper ME, Devereux RB, Dahlof B, Ibsen H, Keane WF, Lindholm LH, Olsen MH, Parving HH, Remuzzi G, Shahinfar S, Snapinn SM, Wachtell K, de Zeeuw D. Renal function and risk for cardiovascular events in type 2 diabetic patients with hypertension: the RENAAL and LIFE studies. J Hypertens. 2007 Apr;25(4):871-6. doi: 10.1097/HJH.0b013e328014953c. PMID 17351381
- [Background] Fossum E, Olsen MH, Hoieggen A, Wachtell K, Reims HM, Kjeldsen SE, Ibsen H, Wan Y, Julius S. Long-term effects of a losartan- compared with an atenolol-based treatment regimen on carotid artery plaque development in hypertensive patients with left ventricular hypertrophy: ICARUS, a LIFE substudy. J Clin Hypertens (Greenwich). 2006 Mar;8(3):169-73. doi: 10.1111/j.1524-6175.2006.04838.x. PMID 16522993
- [Background] Fossum E, Olsen MH, Hoieggen A, Wachtell K, Reims HM, Ibsen H, Julius S, Kjeldsen SE. Long-term plasma catecholamines in patients with hypertension and left ventricular hypertrophy treated with losartan or atenolol: ICARUS, a LIFE substudy. J Hum Hypertens. 2004 Jun;18(6):375-80. doi: 10.1038/sj.jhh.1001712. PMID 15057253
- [Background] Gerdts E, Wachtell K, Omvik P, Otterstad JE, Oikarinen L, Boman K, Dahlof B, Devereux RB. Left atrial size and risk of major cardiovascular events during antihypertensive treatment: losartan intervention for endpoint reduction in hypertension trial. Hypertension. 2007 Feb;49(2):311-6. doi: 10.1161/01.HYP.0000254322.96189.85. Epub 2006 Dec 18. PMID 17178978
- [Background] Gerdts E, Okin PM, de Simone G, Cramariuc D, Wachtell K, Boman K, Devereux RB. Gender differences in left ventricular structure and function during antihypertensive treatment: the Losartan Intervention for Endpoint Reduction in Hypertension Study. Hypertension. 2008 Apr;51(4):1109-14. doi: 10.1161/HYPERTENSIONAHA.107.107474. Epub 2008 Feb 7. PMID 18259011
- [Background] Hildebrandt P, Boesen M, Olsen M, Wachtell K, Groenning B. N-terminal pro brain natriuretic peptide in arterial hypertension--a marker for left ventricular dimensions and prognosis. Eur J Heart Fail. 2004 Mar 15;6(3):313-7. doi: 10.1016/j.ejheart.2004.01.001. PMID 14987582
- [Background] Gerdts E, Papademetriou V, Palmieri V, Boman K, Bjornstad H, Wachtell K, Giles TD, Dahlof B, Devereux RB; Losartan Intervention For End (LIFE) point reduction in hypertension study. Correlates of pulse pressure reduction during antihypertensive treatment (losartan or atenolol) in hypertensive patients with electrocardiographic left ventricular hypertrophy (the LIFE study). Am J Cardiol. 2002 Feb 15;89(4):399-402. doi: 10.1016/s0002-9149(01)02260-3. PMID 11835919
- [Background] Gerdts E, Roman MJ, Palmieri V, Wachtell K, Smith G, Nieminen MS, Dahlof B, Devereux RB. Impact of age on left ventricular hypertrophy regression during antihypertensive treatment with losartan or atenolol (the LIFE study). J Hum Hypertens. 2004 Jun;18(6):417-22. doi: 10.1038/sj.jhh.1001718. PMID 15103312
- [Background] Hoieggen A, Alderman MH, Kjeldsen SE, Julius S, Devereux RB, De Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H, Chen C, Dahlof B; LIFE Study Group. The impact of serum uric acid on cardiovascular outcomes in the LIFE study. Kidney Int. 2004 Mar;65(3):1041-9. doi: 10.1111/j.1523-1755.2004.00484.x. PMID 14871425
- [Background] Gerdts E, Zabalgoitia M, Bjornstad H, Svendsen TL, Devereux RB. Gender differences in systolic left ventricular function in hypertensive patients with electrocardiographic left ventricular hypertrophy (the LIFE study). Am J Cardiol. 2001 Apr 15;87(8):980-3; A4. doi: 10.1016/s0002-9149(01)01433-3. PMID 11305990
- [Background] Ibsen H, Olsen MH, Wachtell K, Borch-Johnsen K, Lindholm LH, Mogensen CE, Dahlof B, Devereux RB, de Faire U, Fyhrquist F, Julius S, Kjeldsen SE, Lederballe-Pedersen O, Nieminen MS, Omvik P, Oparil S, Wan Y. Reduction in albuminuria translates to reduction in cardiovascular events in hypertensive patients: losartan intervention for endpoint reduction in hypertension study. Hypertension. 2005 Feb;45(2):198-202. doi: 10.1161/01.HYP.0000154082.72286.2a. Epub 2005 Jan 17. PMID 15655123
- [Background] Hildebrandt P, Wachtell K, Dahlof B, Papademitriou V, Gerdts E, Giles T, Oikarinen L, Tuxen C, Olsen MH, Devereux RB. Impairment of cardiac function in hypertensive patients with Type 2 diabetes: a LIFE study. Diabet Med. 2005 Aug;22(8):1005-11. doi: 10.1111/j.1464-5491.2005.01564.x. PMID 16026365
- [Background] Ibsen H, Olsen MH, Wachtell K, Borch-Johnsen K, Lindholm LH, Mogensen CE, Dahlof B, Snapinn SM, Wan Y, Lyle PA. Does albuminuria predict cardiovascular outcomes on treatment with losartan versus atenolol in patients with diabetes, hypertension, and left ventricular hypertrophy? The LIFE study. Diabetes Care. 2006 Mar;29(3):595-600. doi: 10.2337/diacare.29.03.06.dc05-1724. PMID 16505512
- [Background] Li ZB, Wachtell K, Okin PM, Gerdts E, Liu JE, Nieminen MS, Jern S, Dahlof B, Devereux RB. Association of left bundle branch block with left ventricular structure and function in hypertensive patients with left ventricular hypertrophy: the LIFE study. J Hum Hypertens. 2004 Jun;18(6):397-402. doi: 10.1038/sj.jhh.1001709. PMID 15071485
- [Background] Oikarinen L, Nieminen MS, Viitasalo M, Toivonen L, Jern S, Dahlof B, Devereux RB, Okin PM; LIFE Study Investigators. QRS duration and QT interval predict mortality in hypertensive patients with left ventricular hypertrophy: the Losartan Intervention for Endpoint Reduction in Hypertension Study. Hypertension. 2004 May;43(5):1029-34. doi: 10.1161/01.HYP.0000125230.46080.c6. Epub 2004 Mar 22. PMID 15037560
- [Background] Julius S, Alderman MH, Beevers G, Dahlof B, Devereux RB, Douglas JG, Edelman JM, Harris KE, Kjeldsen SE, Nesbitt S, Randall OS, Wright JT Jr. Cardiovascular risk reduction in hypertensive black patients with left ventricular hypertrophy: the LIFE study. J Am Coll Cardiol. 2004 Mar 17;43(6):1047-55. doi: 10.1016/j.jacc.2003.11.029. PMID 15028365
- [Background] Kizer JR, Dahlof B, Kjeldsen SE, Julius S, Beevers G, de Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H, Wachtell K, Edelman JM, Snapinn SM, Harris KE, Devereux RB. Stroke reduction in hypertensive adults with cardiac hypertrophy randomized to losartan versus atenolol: the Losartan Intervention For Endpoint reduction in hypertension study. Hypertension. 2005 Jan;45(1):46-52. doi: 10.1161/01.HYP.0000151324.05355.1c. Epub 2004 Dec 6. PMID 15583076
- [Background] McInnes G, Burke TA, Carides G. Cost-effectiveness of losartan-based therapy in patients with hypertension and left ventricular hypertrophy: a UK-based economic evaluation of the Losartan Intervention for Endpoint reduction in hypertension (LIFE) study. J Hum Hypertens. 2006 Jan;20(1):51-8. doi: 10.1038/sj.jhh.1001939. PMID 16357874
- [Background] Kristianson K, Fyhrquist F, Devereux RB, Kjeldsen SE, Lindholm LH, Lyle PA, Nieminen MS, Snapinn SM. An analysis of cholesterol control and statin use in the Losartan Intervention for Endpoint Reduction in Hypertension Study. Clin Ther. 2003 Apr;25(4):1186-99. doi: 10.1016/s0149-2918(03)80075-9. PMID 12809965
- [Background] Okin PM, Devereux RB, Gerdts E, Snapinn SM, Harris KE, Jern S, Kjeldsen SE, Julius S, Edelman JM, Lindholm LH, Dahlof B; LIFE Study Investigators. Impact of diabetes mellitus on regression of electrocardiographic left ventricular hypertrophy and the prediction of outcome during antihypertensive therapy: the Losartan Intervention For Endpoint (LIFE) Reduction in Hypertension Study. Circulation. 2006 Mar 28;113(12):1588-96. doi: 10.1161/CIRCULATIONAHA.105.574822. Epub 2006 Mar 13. PMID 16534012
- [Background] Okin PM, Devereux RB, Nieminen MS, Jern S, Oikarinen L, Viitasalo M, Toivonen L, Kjeldsen SE, Julius S, Dahlof B. Relationship of the electrocardiographic strain pattern to left ventricular structure and function in hypertensive patients: the LIFE study. Losartan Intervention For End point. J Am Coll Cardiol. 2001 Aug;38(2):514-20. doi: 10.1016/s0735-1097(01)01378-x. PMID 11499746
- [Background] Oikarinen L, Nieminen MS, Toivonen L, Viitasalo M, Wachtell K, Papademetriou V, Jern S, Dahlof B, Devereux RB, Okin PM; LIFE Study Investigators. Relation of QT interval and QT dispersion to regression of echocardiographic and electrocardiographic left ventricular hypertrophy in hypertensive patients: the Losartan Intervention For Endpoint Reduction (LIFE) study. Am Heart J. 2003 May;145(5):919-25. doi: 10.1016/S0002-8703(02)94785-X. PMID 12766755
- [Background] Kontos J, Papademetriou V, Wachtell K, Palmieri V, Liu JE, Gerdts E, Boman K, Nieminen MS, Dahlof B, Devereux RB. Impact of valvular regurgitation on left ventricular geometry and function in hypertensive patients with left ventricular hypertrophy: the LIFE study. J Hum Hypertens. 2004 Jun;18(6):431-6. doi: 10.1038/sj.jhh.1001715. PMID 15042117
- [Background] Ibsen H, Wachtell K, Olsen MH, Borch-Johnsen K, Lindholm LH, Mogensen CE, Dahlof B. Albuminuria and cardiovascular risk in hypertensive patients with left ventricular hypertrophy: the LIFE Study. Kidney Int Suppl. 2004 Nov;(92):S56-8. doi: 10.1111/j.1523-1755.2004.09214.x. PMID 15485419
- [Background] Okin PM, Devereux RB, Harris KE, Jern S, Kjeldsen SE, Julius S, Edelman JM, Dahlof B; LIFE Study Investigators. Regression of electrocardiographic left ventricular hypertrophy is associated with less hospitalization for heart failure in hypertensive patients. Ann Intern Med. 2007 Sep 4;147(5):311-9. doi: 10.7326/0003-4819-147-5-200709040-00006. PMID 17785486
- [Background] Okin PM, Devereux RB, Jern S, Julius S, Kjeldsen SE, Dahlof B. Relation of echocardiographic left ventricular mass and hypertrophy to persistent electrocardiographic left ventricular hypertrophy in hypertensive patients: the LIFE Study. Am J Hypertens. 2001 Aug;14(8 Pt 1):775-82. doi: 10.1016/s0895-7061(01)01291-2. PMID 11497193
- [Background] Ibsen H, Olsen MH, Wachtell K, Borch-Johnsen K, Lindholm LH, Mogensen CE. Reduction in albuminuria translates to reduction in cardiovascular events in hypertensive patients with left ventricular hypertrophy and diabetes. J Nephrol. 2008 Jul-Aug;21(4):566-9. PMID 18651547
- [Background] Oikarinen L, Nieminen MS, Viitasalo M, Toivonen L, Wachtell K, Papademetriou V, Jern S, Dahlof B, Devereux RB, Okin PM. Relation of QT interval and QT dispersion to echocardiographic left ventricular hypertrophy and geometric pattern in hypertensive patients. The LIFE study. The Losartan Intervention For Endpoint Reduction. J Hypertens. 2001 Oct;19(10):1883-91. doi: 10.1097/00004872-200110000-00025. PMID 11593111
- [Background] Lindholm LH, Dahlof B, Edelman JM, Ibsen H, Borch-Johnsen K, Olsen MH, Snapinn S, Wachtell K; LIFE study group. Effect of losartan on sudden cardiac death in people with diabetes: data from the LIFE study. Lancet. 2003 Aug 23;362(9384):619-20. doi: 10.1016/S0140-6736(03)14183-9. PMID 12944063
- [Background] Jonsson B, Carides GW, Burke TA, Dasbach EJ, Lindholm LH, Dahlof B; LIFE Study Group. Cost effectiveness of losartan in patients with hypertension and LVH: an economic evaluation for Sweden of the LIFE trial. J Hypertens. 2005 Jul;23(7):1425-31. doi: 10.1097/01.hjh.0000173527.73179.f5. PMID 15942467
- [Background] Okin PM, Devereux RB, Nieminen MS, Jern S, Oikarinen L, Viitasalo M, Toivonen L, Kjeldsen SE, Dahlof B; LIFE Study Investigators. Electrocardiographic strain pattern and prediction of new-onset congestive heart failure in hypertensive patients: the Losartan Intervention for Endpoint Reduction in Hypertension (LIFE) study. Circulation. 2006 Jan 3;113(1):67-73. doi: 10.1161/CIRCULATIONAHA.105.569491. Epub 2005 Dec 19. PMID 16365195
- [Background] Kjeldsen SE, Lyle PA, Kizer JR, Dahlof B, Devereux RB, Julius S, Beevers G, de Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Snapinn SM, Harris KE, Wedel H; LIFE Study Group. The effects of losartan compared to atenolol on stroke in patients with isolated systolic hypertension and left ventricular hypertrophy. The LIFE study. J Clin Hypertens (Greenwich). 2005 Mar;7(3):152-8. doi: 10.1111/j.1524-6175.2005.04254.x. PMID 15785156
- [Background] Okin PM, Devereux RB, Liu JE, Oikarinen L, Jern S, Kjeldsen SE, Julius S, Wachtell K, Nieminen MS, Dahlof B. Regression of electrocardiographic left ventricular hypertrophy predicts regression of echocardiographic left ventricular mass: the LIFE study. J Hum Hypertens. 2004 Jun;18(6):403-9. doi: 10.1038/sj.jhh.1001707. PMID 15057252
- [Background] Narayan P, Papademetriou V, Wachtell K, Gerdts E, Boman K, Nieminen MS, de Simone G, Dahlof B, Fyhrquist F, Hoieggen A, Devereux RB. Association of hemoglobin delivery with left ventricular structure and function in hypertensive patients: Losartan Intervention for End Point Reduction in Hypertension Study. Hypertension. 2006 May;47(5):868-73. doi: 10.1161/01.HYP.0000215578.40687.6f. Epub 2006 Mar 27. PMID 16567586
- [Background] Okin PM, Devereux RB, Jern S, Kjeldsen SE, Julius S, Dahlof B. Baseline characteristics in relation to electrocardiographic left ventricular hypertrophy in hypertensive patients: the Losartan intervention for endpoint reduction (LIFE) in hypertension study. The Life Study Investigators. Hypertension. 2000 Nov;36(5):766-73. doi: 10.1161/01.hyp.36.5.766. PMID 11082141
- [Background] Okin PM, Devereux RB, Jern S, Kjeldsen SE, Julius S, Nieminen MS, Snapinn S, Harris KE, Aurup P, Edelman JM, Wedel H, Lindholm LH, Dahlof B; LIFE Study Investigators. Regression of electrocardiographic left ventricular hypertrophy during antihypertensive treatment and the prediction of major cardiovascular events. JAMA. 2004 Nov 17;292(19):2343-9. doi: 10.1001/jama.292.19.2343. PMID 15547161
- [Background] Kjeldsen SE, Dahlof B, Devereux RB, Julius S, de Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H. Lowering of blood pressure and predictors of response in patients with left ventricular hypertrophy: the LIFE study. Losartan Intervention For Endpoint. Am J Hypertens. 2000 Aug;13(8):899-906. doi: 10.1016/s0895-7061(00)00280-6. PMID 10950398
- [Background] Okin PM, Jern S, Devereux RB, Kjeldsen SE, Dahlof B; LIFE Study Group. Effect of obesity on electrocardiographic left ventricular hypertrophy in hypertensive patients : the losartan intervention for endpoint (LIFE) reduction in hypertension study. Hypertension. 2000 Jan;35(1 Pt 1):13-8. doi: 10.1161/01.hyp.35.1.13. PMID 10642268
- [Background] Olsen MH, Fossum E, Hjerkinn E, Wachtell K, Hoieggen A, Nesbitt SD, Andersen UB, Phillips RA, Gaboury CL, Ibsen H, Kjeldsen SE, Julius S. Relative influence of insulin resistance versus blood pressure on vascular changes in longstanding hypertension. ICARUS, a LIFE sub study. Insulin Carotids US Scandinavia. J Hypertens. 2000 Jan;18(1):75-81. doi: 10.1097/00004872-200018010-00011. PMID 10678546
- [Background] Olsen MH, Andersen UB, Wachtell K, Ibsen H, Dige-Petersen H. Influence of non-steady state during isoglycemic hyperinsulinemic clamp in hypertension. A LIFE substudy. Blood Press. 1999;8(4):207-13. doi: 10.1080/080370599439580. PMID 10697300
- [Background] Olsen MH, Andersen UB, Wachtell K, Ibsen H, Dige-Petersen H. A possible link between endothelial dysfunction and insulin resistance in hypertension. A LIFE substudy. Losartan Intervention For Endpoint-Reduction in Hypertension. Blood Press. 2000;9(2-3):132-9. doi: 10.1080/080370500453474. PMID 10855737
- [Background] Palmieri V, Wachtell K, Gerdts E, Bella JN, Papademetriou V, Tuxen C, Nieminen MS, Dahlof B, de Simone G, Devereux RB. Left ventricular function and hemodynamic features of inappropriate left ventricular hypertrophy in patients with systemic hypertension: the LIFE study. Am Heart J. 2001 May;141(5):784-91. doi: 10.1067/mhj.2001.114803. PMID 11320367
- [Background] Papademetriou V, Devereux RB, Narayan P, Wachtell K, Bella JN, Gerdts E, Chrysant SG, Dahlof B. Similar effects of isolated systolic and combined hypertension on left ventricular geometry and function: the LIFE Study. Am J Hypertens. 2001 Aug;14(8 Pt 1):768-74. doi: 10.1016/s0895-7061(01)01292-4. PMID 11497192
- [Background] Olsen MH, Wachtell K, Aalkjaer C, Devereux RB, Dige-Petersen H, Ibsen H. Endothelial dysfunction in resistance arteries is related to high blood pressure and circulating low density lipoproteins in previously treated hypertension. Am J Hypertens. 2001 Sep;14(9 Pt 1):861-7. doi: 10.1016/s0895-7061(01)02148-3. PMID 11587150
- [Background] Olsen MH, Wachtell K, Hermann KL, Bella JN, Andersen UB, Dige-Petersen H, Rokkedal J, Ibsen H. Maximal exercise capacity is related to cardiovascular structure in patients with longstanding hypertension. A LIFE substudy. Losartan Intervention For Endpoint-Reduction in Hypertension. Am J Hypertens. 2001 Dec;14(12):1205-10. doi: 10.1016/s0895-7061(01)02223-3. PMID 11775128
- [Background] Olsen MH, Wachtell K, Borch-Johnsen K, Okin PM, Kjeldsen SE, Dahlof B, Devereux RB, Ibsen H. A blood pressure independent association between glomerular albumin leakage and electrocardiographic left ventricular hypertrophy. The LIFE Study. Losartan Intervention For Endpoint reduction. J Hum Hypertens. 2002 Aug;16(8):591-5. doi: 10.1038/sj.jhh.1001450. PMID 12149666
- [Background] Okin PM, Wright JT, Nieminen MS, Jern S, Taylor AL, Phillips R, Papademetriou V, Clark LT, Ofili EO, Randall OS, Oikarinen L, Viitasalo M, Toivonen L, Julius S, Dahlof B, Devereux RB. Ethnic differences in electrocardiographic criteria for left ventricular hypertrophy: the LIFE study. Losartan Intervention For Endpoint. Am J Hypertens. 2002 Aug;15(8):663-71. doi: 10.1016/s0895-7061(02)02945-x. PMID 12160187
- [Background] Olsen MH, Wachtell K, Hermann KL, Frandsen E, Dige-Petersen H, Rokkedal J, Devereux RB, Ibsen H. Is cardiovascular remodeling in patients with essential hypertension related to more than high blood pressure? A LIFE substudy. Losartan Intervention For Endpoint-Reduction in Hypertension. Am Heart J. 2002 Sep;144(3):530-7. doi: 10.1067/mhj.2002.124863. PMID 12228792
- [Background] Olsen MH, Wachtell K, Hermann KL, Bella JN, Dige-Petersen H, Rokkedal J, Ibsen H. Left ventricular hypertrophy is associated with reduced vasodilatory capacity in the brachial artery in patients with longstanding hypertension. A LIFE substudy. Blood Press. 2002;11(5):285-92. doi: 10.1080/080370502320779494. PMID 12458651
- [Background] Palmieri V, Okin PM, Bella JN, Gerdts E, Wachtell K, Gardin J, Papademetriou V, Nieminen MS, Dahlof B, Devereux RB; Losartan Intervention For End-point reduction in hypertension. Echocardiographic wall motion abnormalities in hypertensive patients with electrocardiographic left ventricular hypertrophy: the LIFE Study. Hypertension. 2003 Jan;41(1):75-82. doi: 10.1161/01.hyp.0000045081.54784.36. PMID 12511533
- [Background] Palmieri V, Bella JN, Roman MJ, Gerdts E, Papademetriou V, Wachtell K, Nieminen MS, Dahlof B, Devereux RB. Pulse pressure/stroke index and left ventricular geometry and function: the LIFE Study. J Hypertens. 2003 Apr;21(4):781-7. doi: 10.1097/00004872-200304000-00022. PMID 12658025
- [Background] Palmieri V, Wachtell K, Bella JN, Gerdts E, Papademetriou V, Nieminen MS, Dahlof B, Roman MJ, Devereux RB. Usefulness of the assessment of the appropriateness of left ventricular mass to detect left ventricular systolic and diastolic abnormalities in absence of echocardiographic left ventricular hypertrophy: the LIFE study. J Hum Hypertens. 2004 Jun;18(6):423-30. doi: 10.1038/sj.jhh.1001719. PMID 15002006
- [Background] Olsen MH, Wachtell K, de Simone G, Palmieri V, Dige-Petersen H, Devereux RB, Ibsen H, Rokkedal J. Is inappropriate left ventricular mass related to neurohormonal factors and/or arterial changes in hypertension? A LIFE substudy. J Hum Hypertens. 2004 Jun;18(6):437-43. doi: 10.1038/sj.jhh.1001720. PMID 15014540
- [Background] Olsen MH, Wachtell K, Bella JN, Palmieri V, Gerdts E, Smith G, Nieminen MS, Dahlof B, Ibsen H, Devereux RB. Albuminuria predicts cardiovascular events independently of left ventricular mass in hypertension: a LIFE substudy. J Hum Hypertens. 2004 Jun;18(6):453-9. doi: 10.1038/sj.jhh.1001711. PMID 15085167
- [Background] Reims HM, Kjeldsen SE, Brady WE, Dahlof B, Devereux RB, Julius S, Beevers G, De Faire U, Fyhrquist F, Ibsen H, Kristianson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H. Alcohol consumption and cardiovascular risk in hypertensives with left ventricular hypertrophy: the LIFE study. J Hum Hypertens. 2004 Jun;18(6):381-9. doi: 10.1038/sj.jhh.1001731. PMID 15103313
- [Background] Okin PM, Devereux RB, Nieminen MS, Jern S, Oikarinen L, Viitasalo M, Toivonen L, Kjeldsen SE, Julius S, Snapinn S, Dahlof B; LIFE Study Investigators. Electrocardiographic strain pattern and prediction of cardiovascular morbidity and mortality in hypertensive patients. Hypertension. 2004 Jul;44(1):48-54. doi: 10.1161/01.HYP.0000132556.91792.6a. Epub 2004 Jun 1. PMID 15173125
- [Background] Olsen MH, Wachtell K, Tuxen C, Fossum E, Bang LE, Hall C, Ibsen H, Rokkedal J, Devereux RB, Hildebrandt P. N-terminal pro-brain natriuretic peptide predicts cardiovascular events in patients with hypertension and left ventricular hypertrophy: a LIFE study. J Hypertens. 2004 Aug;22(8):1597-604. doi: 10.1097/01.hjh.0000125451.28861.2a. PMID 15257184
- [Background] Olsen MH, Wachtell K, Bella JN, Liu JE, Boman K, Gerdts E, Papademetriou V, Nieminen MS, Rokkedal J, Dahlof B, Devereux RB. Effect of losartan versus atenolol on aortic valve sclerosis (a LIFE substudy). Am J Cardiol. 2004 Oct 15;94(8):1076-80. doi: 10.1016/j.amjcard.2004.06.074. PMID 15476632
- [Background] Olsen MH, Wachtell K, Bella JN, Gerdts E, Palmieri V, Nieminen MS, Smith G, Ibsen H, Devereux RB; LIFE substudy. Aortic valve sclerosis relates to cardiovascular events in patients with hypertension (a LIFE substudy). Am J Cardiol. 2005 Jan 1;95(1):132-6. doi: 10.1016/j.amjcard.2004.08.080. PMID 15619412
- [Background] Olsen MH, Christensen MK, Wachtell K, Tuxen C, Fossum E, Bang LE, Wiinberg N, Devereux RB, Kjeldsen SE, Hildebrandt P, Dige-Petersen H, Rokkedal J, Ibsen H. Markers of collagen synthesis is related to blood pressure and vascular hypertrophy: a LIFE substudy. J Hum Hypertens. 2005 Apr;19(4):301-7. doi: 10.1038/sj.jhh.1001819. PMID 15647776
- [Background] Reims HM, Oparil S, Kjeldsen SE, Devereux RB, Julius S, Brady WE, Fyhrquist F, Ibsen H, Lindholm LH, Omvik P, Wedel H, Beevers G, de Faire U, Kristianson K, Lederballe-Pedersen O, Nieminen MS, Dahlof B; LIFE Study Group. Losartan benefits over atenolol in non-smoking hypertensive patients with left ventricular hypertrophy: the LIFE study. Blood Press. 2004;13(6):376-84. doi: 10.1080/08037050410016483. PMID 15771223
- [Background] Olsen MH, Fossum E, Hoieggen A, Wachtell K, Hjerkinn E, Nesbitt SD, Andersen UB, Phillips RA, Gaboury CL, Ibsen H, Kjeldsen SE, Julius S. Long-term treatment with losartan versus atenolol improves insulin sensitivity in hypertension: ICARUS, a LIFE substudy. J Hypertens. 2005 Apr;23(4):891-8. doi: 10.1097/01.hjh.0000163160.60234.15. PMID 15775796
- [Background] Olsen MH, Wachtell K, Tuxen C, Fossum E, Bang LE, Hall C, Ibsen H, Rokkedal J, Devereux RB, Hildebrandt PR. Opposite effects of losartan and atenolol on natriuretic peptides in patients with hypertension and left ventricular hypertrophy: a LIFE substudy. J Hypertens. 2005 May;23(5):1083-90. doi: 10.1097/01.hjh.0000166851.18463.85. PMID 15834296
- [Background] Olsen MH, Wachtell K, Neland K, Bella JN, Rokkedal J, Dige-Petersen H, Ibsen H. Losartan but not atenolol reduce carotid artery hypertrophy in essential hypertension. A LIFE substudy. Blood Press. 2005;14(3):177-83. doi: 10.1080/08037050510034185. PMID 16036498
- [Background] Olsen MH, Wachtell K, Bella JN, Palmieri V, Gerdts E, Smith G, Nieminen MS, Dahlof B, Ibsen H, Devereux RB. Aortic valve sclerosis and albuminuria predict cardiovascular events independently in hypertension: a losartan intervention for endpoint-reduction in hypertension (LIFE) substudy. Am J Hypertens. 2005 Nov;18(11):1430-6. doi: 10.1016/j.amjhyper.2005.05.030. PMID 16280277
- [Background] Olsen MH, Wachtell K, Ibsen H, Lindholm LH, Dahlof B, Devereux RB, Kjeldsen SE, Oikarinen L, Okin PM; LIFE Study Investigators. Reductions in albuminuria and in electrocardiographic left ventricular hypertrophy independently improve prognosis in hypertension: the LIFE study. J Hypertens. 2006 Apr;24(4):775-81. doi: 10.1097/01.hjh.0000217862.50735.dc. PMID 16531808
- [Background] Olsen MH, Wachtell K, Dahlof B, Devereux RB, Ibsen H, Kjeldsen SE, Lindholm LH, Lyle PA, Nieminen MS. The effect of losartan compared with atenolol on the incidence of revascularization in patients with hypertension and electrocardiographic left ventricular hypertrophy. The LIFE study. J Hum Hypertens. 2006 Jun;20(6):460-4. doi: 10.1038/sj.jhh.1002013. No abstract available. PMID 16572193
- [Background] Palmieri V, Okin PM, de Simone G, Bella JN, Wachtell K, Gerdts E, Boman K, Nieminen MS, Dahlof B, Devereux RB. Electrocardiographic characteristics and metabolic risk factors associated with inappropriately high left ventricular mass in patients with electrocardiographic left ventricular hypertrophy: the LIFE Study. J Hypertens. 2007 May;25(5):1079-85. doi: 10.1097/HJH.0b013e3280825638. PMID 17414673
- [Background] Okin PM, Wachtell K, Devereux RB, Nieminen MS, Oikarinen L, Viitasalo M, Toivonen L, Ibsen H, Olsen MH, Borch-Johnsen K, Lindholm LH, Kjeldsen SE, Julius S, Dahlof B; LIFE Study Investigators. Combination of the electrocardiographic strain pattern and albuminuria for the prediction of new-onset heart failure in hypertensive patients: the LIFE study. Am J Hypertens. 2008 Mar;21(3):273-9. doi: 10.1038/ajh.2007.66. Epub 2008 Jan 24. PMID 18219298
- [Background] Palmieri V, Bella JN, Gerdts E, Wachtell K, Papademetriou V, Nieminen MS, Dahlof B, Devereux RB. Change in pulse pressure/stroke index in response to sustained blood pressure reduction and its impact on left ventricular mass and geometry changes: the life study. Am J Hypertens. 2008 Jun;21(6):701-7. doi: 10.1038/ajh.2008.162. Epub 2008 Apr 10. PMID 18437127
- [Background] Wachtell K, Bella JN, Liebson PR, Gerdts E, Dahlof B, Aalto T, Roman MJ, Papademetriou V, Ibsen H, Rokkedal J, Devereux RB. Impact of different partition values on prevalences of left ventricular hypertrophy and concentric geometry in a large hypertensive population : the LIFE study. Hypertension. 2000 Jan;35(1 Pt 1):6-12. doi: 10.1161/01.hyp.35.1.6. PMID 10642267
- [Background] Hoieggen A, Fossum E, Nesbitt SD, Palmieri V, Kjeldsen SE. Blood viscosity, plasma adrenaline and fasting insulin in hypertensive patients with left ventricular hypertrophy. ICARUS, a LIFE Substudy. Insulin CARotids US Scandinavica. Blood Press. 2000;9(2-3):83-90. doi: 10.1080/08037050050151771. PMID 10855729
- [Background] Wachtell K, Rokkedal J, Bella JN, Aalto T, Dahlof B, Smith G, Roman MJ, Ibsen H, Aurigemma GP, Devereux RB. Effect of electrocardiographic left ventricular hypertrophy on left ventricular systolic function in systemic hypertension (The LIFE Study). Losartan Intervention For Endpoint. Am J Cardiol. 2001 Jan 1;87(1):54-60. doi: 10.1016/s0002-9149(00)01272-8. PMID 11137834
- [Background] Zabalgoitia M, Berning J, Koren MJ, Stoylen A, Nieminen MS, Dahlof B, Devereux RB; LIFE Study Investigators. Impact of coronary artery disease on left ventricular systolic function and geometry in hypertensive patients with left ventricular hypertrophy (the LIFE study). Am J Cardiol. 2001 Sep 15;88(6):646-50. doi: 10.1016/s0002-9149(01)01807-0. PMID 11564388
- [Background] Wachtell K, Palmieri V, Olsen MH, Bella JN, Aalto T, Dahlof B, Gerdts E, Wright JT Jr, Papademetriou V, Mogensen CE, Borch-Johnsen K, Ibsen H, Devereux RB. Urine albumin/creatinine ratio and echocardiographic left ventricular structure and function in hypertensive patients with electrocardiographic left ventricular hypertrophy: the LIFE study. Losartan Intervention for Endpoint Reduction. Am Heart J. 2002 Feb;143(2):319-26. doi: 10.1067/mhj.2002.119895. PMID 11835038
- [Background] Wachtell K, Olsen MH, Dahlof B, Devereux RB, Kjeldsen SE, Nieminen MS, Okin PM, Papademetriou V, Mogensen CE, Borch-Johnsen K, Ibsen H. Microalbuminuria in hypertensive patients with electrocardiographic left ventricular hypertrophy: the LIFE study. J Hypertens. 2002 Mar;20(3):405-12. doi: 10.1097/00004872-200203000-00015. PMID 11875307
- [Background] Wachtell K, Bella JN, Rokkedal J, Palmieri V, Papademetriou V, Dahlof B, Aalto T, Gerdts E, Devereux RB. Change in diastolic left ventricular filling after one year of antihypertensive treatment: The Losartan Intervention For Endpoint Reduction in Hypertension (LIFE) Study. Circulation. 2002 Mar 5;105(9):1071-6. doi: 10.1161/hc0902.104599. PMID 11877357
- [Background] Wachtell K, Palmieri V, Olsen MH, Gerdts E, Papademetriou V, Nieminen MS, Smith G, Dahlof B, Aurigemma GP, Devereux RB. Change in systolic left ventricular performance after 3 years of antihypertensive treatment: the Losartan Intervention for Endpoint (LIFE) Study. Circulation. 2002 Jul 9;106(2):227-32. doi: 10.1161/01.cir.0000021601.49664.2a. PMID 12105163
- [Background] Wachtell K, Dahlof B, Rokkedal J, Papademetriou V, Nieminen MS, Smith G, Gerdts E, Boman K, Bella JN, Devereux RB. Change of left ventricular geometric pattern after 1 year of antihypertensive treatment: the Losartan Intervention For Endpoint reduction in hypertension (LIFE) study. Am Heart J. 2002 Dec;144(6):1057-64. doi: 10.1067/mhj.2002.126113. PMID 12486431
- [Background] Wachtell K, Ibsen H, Olsen MH, Borch-Johnsen K, Lindholm LH, Mogensen CE, Dahlof B, Devereux RB, Beevers G, de Faire U, Fyhrquist F, Julius S, Kjeldsen SE, Kristianson K, Lederballe-Pedersen O, Nieminen MS, Okin PM, Omvik P, Oparil S, Wedel H, Snapinn SM, Aurup P. Albuminuria and cardiovascular risk in hypertensive patients with left ventricular hypertrophy: the LIFE study. Ann Intern Med. 2003 Dec 2;139(11):901-6. doi: 10.7326/0003-4819-139-11-200312020-00008. PMID 14644892
- [Background] Wiinberg N, Bang LE, Wachtell K, Larsen J, Olsen MH, Tuxen C, Hildebrandt PR, Rokkedal J, Ibsen H, Devereux RB. 24-h Ambulatory blood pressure in patients with ECG-determined left ventricular hypertrophy: left ventricular geometry and urinary albumin excretion-a LIFE substudy. J Hum Hypertens. 2004 Jun;18(6):391-6. doi: 10.1038/sj.jhh.1001717. PMID 15057254
- [Background] Wachtell K, Papademetriou V, Smith G, Gerdts E, Dahlof B, Engblom E, Aurigemma GP, Bella JN, Ibsen H, Rokkedal J, Devereux RB. Relation of impaired left ventricular filling to systolic midwall mechanics in hypertensive patients with normal left ventricular systolic chamber function: the Losartan Intervention for Endpoint Reduction in Hypertension (LIFE) study. Am Heart J. 2004 Sep;148(3):538-44. doi: 10.1016/j.ahj.2004.03.015. PMID 15389245
- [Background] Dahlof B, Devereux RB, Kjeldsen SE, Lyle PA, Zhang Z, Edelman JM. Atenolol as a comparator in outcome trials in hypertension: a correct choice in the past, but not for the future? Blood Press. 2007;16(1):6-12. doi: 10.1080/08037050701246386. PMID 17453746
- [Background] de Simone G, Olsen MH, Wachtell K, Hille DA, Dahlof B, Ibsen H, Kjeldsen SE, Lyle PA, Devereux RB. Clusters of metabolic risk factors predict cardiovascular events in hypertension with target-organ damage: the LIFE study. J Hum Hypertens. 2007 Aug;21(8):625-32. doi: 10.1038/sj.jhh.1002203. Epub 2007 May 3. PMID 17476291
- [Background] Wachtell K, Okin PM, Olsen MH, Dahlof B, Devereux RB, Ibsen H, Kjeldsen SE, Lindholm LH, Nieminen MS, Thygesen K. Regression of electrocardiographic left ventricular hypertrophy during antihypertensive therapy and reduction in sudden cardiac death: the LIFE Study. Circulation. 2007 Aug 14;116(7):700-5. doi: 10.1161/CIRCULATIONAHA.106.666594. Epub 2007 Jul 30. PMID 17664372
- [Background] Smebye ML, Iversen EK, Hoieggen A, Flaa A, Os I, Kjeldsen SE, Olsen MH, Chattopadhyay A, Hille DA, Lyle PA, Devereux RB, Dahlof B. Effect of hemoglobin levels on cardiovascular outcomes in patients with isolated systolic hypertension and left ventricular hypertrophy (from the LIFE study). Am J Cardiol. 2007 Sep 1;100(5):855-9. doi: 10.1016/j.amjcard.2007.03.109. Epub 2007 Jul 2. PMID 17719333
- [Background] Okin PM, Devereux RB, Harris KE, Jern S, Kjeldsen SE, Lindholm LH, Dahlof B; LIFE Study Investigators. In-treatment resolution or absence of electrocardiographic left ventricular hypertrophy is associated with decreased incidence of new-onset diabetes mellitus in hypertensive patients: the Losartan Intervention for Endpoint Reduction in Hypertension (LIFE) Study. Hypertension. 2007 Nov;50(5):984-90. doi: 10.1161/HYPERTENSIONAHA.107.096818. Epub 2007 Sep 24. PMID 17893425
- [Background] Os I, Franco V, Kjeldsen SE, Manhem K, Devereux RB, Gerdts E, Hille DA, Lyle PA, Okin PM, Dahlof B, Oparil S. Effects of losartan in women with hypertension and left ventricular hypertrophy: results from the Losartan Intervention for Endpoint Reduction in Hypertension Study. Hypertension. 2008 Apr;51(4):1103-8. doi: 10.1161/HYPERTENSIONAHA.107.105296. Epub 2008 Feb 7. PMID 18259029
- [Background] Cicala S, de Simone G, Wachtell K, Gerdts E, Boman K, Nieminen MS, Dahlof B, Devereux RB. Clinical impact of 'in-treatment' wall motion abnormalities in hypertensive patients with left ventricular hypertrophy: the LIFE study. J Hypertens. 2008 Apr;26(4):806-12. doi: 10.1097/HJH.0b013e3282f4b3a9. PMID 18327092
- [Background] Olsen MH, Wachtell K, Beevers G, Dahlof B, de Simone G, Devereux RB, de Faire U, Fyhrquist F, Ibsen H, Kjeldsen SE, Lederballe-Pedersen O, Lindholm LH, Lyle PA, Nieminen MS, Omvik P, Oparil S, Wedel H. Effects of losartan compared with atenolol on lipids in patients with hypertension and left ventricular hypertrophy: the Losartan Intervention For Endpoint reduction in hypertension study. J Hypertens. 2009 Mar;27(3):567-74. doi: 10.1097/HJH.0b013e32831daf96. PMID 19262226
- [Background] Gerdts E, Okin PM, Omvik P, Wachtell K, Dahlof B, Hildebrandt P, Nieminen MS, Devereux RB. Impact of diabetes on treatment-induced changes in left ventricular structure and function in hypertensive patients with left ventricular hypertrophy. The LIFE study. Nutr Metab Cardiovasc Dis. 2009 Jun;19(5):306-12. doi: 10.1016/j.numecd.2008.12.009. Epub 2009 Mar 19. PMID 19303268
- [Background] Olsen MH, Wachtell K, Beevers G, Dahlof B, Devereux RB, de Faire U, Fyhrquist F, Ibsen H, Kjeldsen SE, Lederballe-Pedersen O, Lindholm LH, Narayan P, Nieminen MS, Omvik P, Oparil S, Wedel H. Prognostic importance of hemoglobin in hypertensive patients with electrocardiographic left ventricular hypertrophy: the Losartan Intervention For End point reduction in hypertension (LIFE) study. Am Heart J. 2009 Jan;157(1):177-84. doi: 10.1016/j.ahj.2008.08.011. Epub 2008 Oct 17. PMID 19081416
- [Background] Boman K, Gerdts E, Wachtell K, Dahlof B, Nieminen MS, Olofsson M, Papademetriou V, Devereux RB. Exercise and cardiovascular outcomes in hypertensive patients in relation to structure and function of left ventricular hypertrophy: the LIFE study. Eur J Cardiovasc Prev Rehabil. 2009 Apr;16(2):242-8. doi: 10.1097/HJR.0b013e328329560e. PMID 19369828
- [Derived] Lilja-Cyron A, Bang CN, Gerdts E, Larstorp AC, Kjeldsen SE, Julius S, Okin PM, Wachtell K, Devereux RB. Aortic Root Dilatation in Hypertensive Patients with Left Ventricular Hypertrophy-Application of A New Multivariate Predictive Model. The Life Study. Rev Cardiovasc Med. 2022 Mar 10;23(3):95. doi: 10.31083/j.rcm2303095. PMID 35345262
- [Derived] Nuotio ML, Sanez Tahtisalo H, Lahtinen A, Donner K, Fyhrquist F, Perola M, Kontula KK, Hiltunen TP. Pharmacoepigenetics of hypertension: genome-wide methylation analysis of responsiveness to four classes of antihypertensive drugs using a double-blind crossover study design. Epigenetics. 2022 Nov;17(11):1432-1445. doi: 10.1080/15592294.2022.2038418. Epub 2022 Feb 25. PMID 35213289
- [Derived] Mengozzi A, Trico D, Natali A. A novel method for interpreting survival analysis data: description and test on three major clinical trials on cardiovascular prevention. Trials. 2020 Jun 26;21(1):578. doi: 10.1186/s13063-020-04511-y. PMID 32586346
- [Derived] Okin PM, Hille DA, Wachtell K, Kjeldsen SE, Julius S, Devereux RB. On-treatment HDL cholesterol predicts incident atrial fibrillation in hypertensive patients with left ventricular hypertrophy. Blood Press. 2020 Oct;29(5):319-326. doi: 10.1080/08037051.2020.1782171. Epub 2020 Jun 25. PMID 32586143
- [Derived] Okin PM, Kjeldsen SE, Devereux RB. Effect of antihypertensive therapy on development of incident conduction system disease in hypertensive patients. J Hypertens. 2019 Mar;37(3):629-635. doi: 10.1097/HJH.0000000000001915. PMID 30676480
- [Derived] Ala-Mutka EM, Rimpela JM, Fyhrquist F, Kontula KK, Hiltunen TP. Effect of hydrochlorothiazide on serum uric acid concentration: a genome-wide association study. Pharmacogenomics. 2018 Apr;19(6):517-527. doi: 10.2217/pgs-2017-0184. Epub 2018 Mar 27. PMID 29580174
- [Derived] Okin PM, Kjeldsen SE, Devereux RB. Impact of achieved systolic blood pressure on renal function in hypertensive patients. Eur Heart J Qual Care Clin Outcomes. 2016 Oct 1;2(4):271-276. doi: 10.1093/ehjqcco/qcw017. PMID 29474712
- [Derived] Okin PM, Kjeldsen SE, Devereux RB. The relationship of all-cause mortality to average on-treatment systolic blood pressure is significantly related to baseline systolic blood pressure: implications for interpretation of the Systolic Blood Pressure Intervention Trial study. J Hypertens. 2018 Apr;36(4):916-923. doi: 10.1097/HJH.0000000000001620. PMID 29176391
- [Derived] Okin PM, Hille DA, Kjeldsen SE, Devereux RB. Combining ECG Criteria for Left Ventricular Hypertrophy Improves Risk Prediction in Patients With Hypertension. J Am Heart Assoc. 2017 Nov 18;6(11):e007564. doi: 10.1161/JAHA.117.007564. PMID 29151037
- [Derived] Vishram JK, Dahlof B, Devereux RB, Ibsen H, Kjeldsen SE, Lindholm LH, Mancia G, Okin PM, Rothwell PM, Wachtell K, Olsen MH. Blood pressure variability predicts cardiovascular events independently of traditional cardiovascular risk factors and target organ damage: a LIFE substudy. J Hypertens. 2015 Dec;33(12):2422-30. doi: 10.1097/HJH.0000000000000739. PMID 26378687
- [Derived] Okin PM, Kjeldsen SE, Devereux RB. Systolic Blood Pressure Control and Mortality After Stroke in Hypertensive Patients. Stroke. 2015 Aug;46(8):2113-8. doi: 10.1161/STROKEAHA.115.009592. Epub 2015 Jun 18. PMID 26089332
- [Derived] Okin PM, Hille DA, Larstorp AC, Wachtell K, Kjeldsen SE, Dahlof B, Devereux RB. Effect of lower on-treatment systolic blood pressure on the risk of atrial fibrillation in hypertensive patients. Hypertension. 2015 Aug;66(2):368-73. doi: 10.1161/HYPERTENSIONAHA.115.05728. Epub 2015 Jun 8. PMID 26056336
- [Derived] Okin PM, Wachtell K, Gerdts E, Dahlof B, Devereux RB. Relationship of left ventricular systolic function to persistence or development of electrocardiographic left ventricular hypertrophy in hypertensive patients: implications for the development of new heart failure. J Hypertens. 2014 Dec;32(12):2472-8; discussion 2478. doi: 10.1097/HJH.0000000000000432. PMID 25340854
- [Derived] Bang CN, Gerdts E, Aurigemma GP, Boman K, de Simone G, Dahlof B, Kober L, Wachtell K, Devereux RB. Four-group classification of left ventricular hypertrophy based on ventricular concentricity and dilatation identifies a low-risk subset of eccentric hypertrophy in hypertensive patients. Circ Cardiovasc Imaging. 2014 May;7(3):422-9. doi: 10.1161/CIRCIMAGING.113.001275. Epub 2014 Apr 10. PMID 24723582
- [Derived] Bang CN, Okin PM, Kober L, Wachtell K, Gottlieb AB, Devereux RB. Psoriasis is associated with subsequent atrial fibrillation in hypertensive patients with left ventricular hypertrophy: the Losartan Intervention For Endpoint study. J Hypertens. 2014 Mar;32(3):667-72. doi: 10.1097/HJH.0000000000000078. PMID 24379001
- [Derived] Okin PM, Bang CN, Wachtell K, Hille DA, Kjeldsen SE, Dahlof B, Devereux RB. Relationship of sudden cardiac death to new-onset atrial fibrillation in hypertensive patients with left ventricular hypertrophy. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):243-51. doi: 10.1161/CIRCEP.112.977777. Epub 2013 Feb 12. PMID 23403268
- [Derived] Larstorp AC, Ariansen I, Gjesdal K, Olsen MH, Ibsen H, Devereux RB, Okin PM, Dahlof B, Kjeldsen SE, Wachtell K. Association of pulse pressure with new-onset atrial fibrillation in patients with hypertension and left ventricular hypertrophy: the Losartan Intervention For Endpoint (LIFE) reduction in hypertension study. Hypertension. 2012 Aug;60(2):347-53. doi: 10.1161/HYPERTENSIONAHA.112.195032. Epub 2012 Jul 2. PMID 22753219
- [Derived] Greve AM, Olsen MH, Bella JN, Lonnebakken MT, Gerdts E, Okin PM, Palmieri V, Boman K, Nieminen MS, Omvik P, Dahlof B, Devereux RB, Wachtell K. Contrasting hemodynamic mechanisms of losartan- vs. atenolol-based antihypertensive treatment: a LIFE study. Am J Hypertens. 2012 Sep;25(9):1017-23. doi: 10.1038/ajh.2012.81. Epub 2012 Jun 14. PMID 22695506
- [Derived] Okin PM, Kjeldsen SE, Lindholm LH, Dahlof B, Devereux RB. The relationship of electrocardiographic left ventricular hypertrophy to decreased serum potassium. Blood Press. 2012 Jun;21(3):146-52. doi: 10.3109/08037051.2011.649537. Epub 2012 Jan 16. PMID 22243363
- [Derived] Lonnebakken MT, Gerdts E, Boman K, Wachtell K, Dahlof B, Devereux RB. In-treatment stroke volume predicts cardiovascular risk in hypertension. J Hypertens. 2011 Aug;29(8):1508-14. doi: 10.1097/HJH.0b013e32834921fb. PMID 21720264
- [Derived] Olsen MH, Wachtell K, Ibsen H, Lindholm L, Kjeldsen SE, Omvik P, Nieminen MS, Dahlof B, Okin PM, Devereux RB. Changes in subclinical organ damage vs. in Framingham risk score for assessing cardiovascular risk reduction during continued antihypertensive treatment: a LIFE substudy. J Hypertens. 2011 May;29(5):997-1004. doi: 10.1097/HJH.0b013e328344daa3. PMID 21358415
- [Derived] Okin PM, Kjeldsen SE, Dahlof B, Devereux RB. Racial differences in incident heart failure during antihypertensive therapy. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):157-64. doi: 10.1161/CIRCOUTCOMES.110.960112. Epub 2011 Feb 8. PMID 21304095
- [Derived] Okin PM, Oikarinen L, Viitasalo M, Toivonen L, Kjeldsen SE, Nieminen MS, Edelman JM, Dahlof B, Devereux RB; LIFE Study Investigators. Serial assessment of the electrocardiographic strain pattern for prediction of new-onset heart failure during antihypertensive treatment: the LIFE study. Eur J Heart Fail. 2011 Apr;13(4):384-91. doi: 10.1093/eurjhf/hfq224. Epub 2011 Jan 14. PMID 21239405
- [Derived] Okin PM, Kjeldsen SE, Julius S, Hille DA, Dahlof B, Edelman JM, Devereux RB. All-cause and cardiovascular mortality in relation to changing heart rate during treatment of hypertensive patients with electrocardiographic left ventricular hypertrophy. Eur Heart J. 2010 Sep;31(18):2271-9. doi: 10.1093/eurheartj/ehq225. Epub 2010 Jul 2. PMID 20601389
- [Derived] Okin PM, Gerdts E, Wachtell K, Oikarinen L, Nieminen MS, Dahlof B, Devereux RB. Relationship of left atrial enlargement to persistence or development of ECG left ventricular hypertrophy in hypertensive patients: implications for the development of new atrial fibrillation. J Hypertens. 2010 Jul;28(7):1534-40. doi: 10.1097/hjh.0b013e328338c20e. PMID 20589977
- [Derived] Kjeldsen SE, Devereux RB, Hille DA, Lyle PA, Dahlof B, Julius S, Edelman JM, Snapinn SM, de Faire U, Fyhrquist F, Ibsen H, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H. Predictors of cardiovascular events in patients with hypertension and left ventricular hypertrophy: the Losartan Intervention for Endpoint reduction in hypertension study. Blood Press. 2009;18(6):348-61. doi: 10.3109/08037050903460590. PMID 20001655
- [Derived] Okin PM, Oikarinen L, Viitasalo M, Toivonen L, Kjeldsen SE, Nieminen MS, Edelman JM, Dahlof B, Devereux RB; LIFE Study Investigators. Prognostic value of changes in the electrocardiographic strain pattern during antihypertensive treatment: the Losartan Intervention for End-Point Reduction in Hypertension Study (LIFE). Circulation. 2009 Apr 14;119(14):1883-91. doi: 10.1161/CIRCULATIONAHA.108.812313. Epub 2009 Mar 30. PMID 19332468